CLINICAL TRIAL: NCT02277925
Title: Permanent Versus Delayed-absorbable Monofilament Suture for Vaginal Graft Attachment During Minimally-invasive Total Hysterectomy and Sacrocolpopexy: A Randomized Clinical Trial
Brief Title: Permanent Versus Absorbable Colpopexy Trial
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Northwestern University (Other); Augusta University (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-2402
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Vaginal mesh exposure rates; Vaginal suture exposure rates
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Polytetrafluoroethylene; Polydioxanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gore-Tex permanent suture (Active Comparator): Participants in this arm will receive Gore-Tex permanent suture
  Interventions: Other: Polytetrafluoroethylene
- PDS delayed absorbable suture (Experimental): Participants in this arm will receive 2-0 PDS delayed absorbable suture
  Interventions: Other: Polydioxanone

INTERVENTIONS:
Other: Polytetrafluoroethylene — Suture used to attach mesh during sacral colpopexy surgery
  Other Names: Gore-Tex permanent suture
  Arms: Gore-Tex permanent suture
Other: Polydioxanone — Suture used to attach mesh during sacral colpopexy surgery
  Other Names: 2-0 PDS delayed absorbable monofilament suture
  Arms: PDS delayed absorbable suture

SUMMARY:
Primary Aim:

The primary aim of this randomized controlled trial (RCT) is to compare vaginal mesh and suture exposure rates in women undergoing robotic total hysterectomy and sacrocolpopexy with a light-weight polypropylene mesh (Upsylon™ y-mesh) using permanent (polytetrafluoroethylene, Gore-Tex) versus delayed absorbable monofilament (2-0 polydioxanone, PDS) sutures through 1-year.

Secondary Aims:

1. To compare the 1-year composite success rate (leading edge of prolapse is at or above the hymen and apex has descended less than 1/3 of the vaginal length, no subjective feeling of bulge; and no retreatment for pelvic organ prolapse (POP) or vaginal mesh exposure) of permanent versus delayed absorbable sutures for mesh graft attachment during robotic total hysterectomy and sacrocolpopexy.
2. To evaluate adverse outcomes in each group

DETAILED DESCRIPTION:
Symptomatic pelvic organ prolapse is common and 13%1 to 19%2,3 of women undergo surgical repair. Reconstructive pelvic surgery is broadly divided into procedures that rely on existing native tissue versus the use of graft augmentation, either with synthetic or biologic materials. Native tissue vaginal repair, while associated with the lowest rate of surgical complications,4 has a high rate of recurrent prolapse. A recent randomized trial of uterosacral versus sacrospinous ligament fixation for POP demonstrated a 30% recurrence rate at 2 years.3

Abdominal sacrocolpopexy (SCP) is considered to be the most durable operation for advanced pelvic organ prolapse with reoperation rates of less than 5%.5-7 Minimally-invasive techniques of SCP, such as robotic-assistance, are associated with improved recovery times and less cost than abdominal SCP without a demonstrable difference in efficacy.8,9 While traditionally reserved for women with vaginal vault prolapse, SCP is increasingly considered as a primary surgical option for women who present with uterovaginal prolapse in an attempt to improve longer-term surgical outcomes. The optimal management of the uterus and cervix in these cases is unclear.

Rationale for total versus supracervical hysterectomy with concomitant SCP

While supracervical hysterectomy and concomitant SCP are associated with lower rates of mesh exposure,10-12 potential negative consequences of a supracervical hysterectomy include morcellation of unanticipated uterine malignancy,13 cervical stump prolapse/elongation, cyclic vaginal bleeding, and reduced anterior vaginal support (Myers EM, Matthews et al., in press). When conducting a supracervical hysterectomy, power morcellators are the most common method used to extract the amputated uterine corpus. The potential risks of power morcellation were recently highlighted by the FDA safety notification which focused on the potential to disseminate fragments of an undiagnosed uterine leiomyosarcoma throughout the abdomen, which negatively impacts prognosis (http://www.fda.gov/MedicalDevices/Safety/AlertsandNotices/ucm393576.htm). With these recent developments the focus has shifted towards performing total hysterectomy for delivery of an intact specimen through the vagina.

Vaginal mesh exposure has been a problematic complication with both abdominal SCP and minimally invasive SCP. Widely disparate rates of mesh exposure ranging from 0%14 to 27%15 have been reported. A systematic review of ASCP outcomes in 2004 reported an overall rate of 3.4%,6 and a recent meta-analysis of robotic-assisted SCP reported an overall rate of 2%.16 Some consistent risk factors for mesh exposure are non-Type 1 polypropylene mesh (knitted, small-pore mesh materials) and smoking.17,18 Some studies have identified total hysterectomy as a significant risk factor. In an evaluation of patients enrolled in the CARE trial, 6% had evidence of mesh exposure at 2 years, with concomitant hysterectomy presenting almost a 5-fold increased risk.18 The rate at 6 years rose to 10.5%. 5 More than 50% of subjects in this trial, however, had a non-Type 1 polypropylene mesh. Akyol et al. demonstrated a 2-fold increased risk (12%)19 and Bensinger et al. a 7-fold increased risk (8.2%)20 of concomitant total hysterectomy. In contrast, 4 retrospective studies in which Type1 polypropylene mesh was used revealed no increased risk of mesh erosion with concomitant total hysterectomy.14,21-23 These widely discrepant rates of mesh exposure may be related to surgical technique, graft material and/or suture materials used for mesh attachment.

Rationale for need to study suture material for mesh attachment during SCP

The effect of suture on mesh exposure may be as significant as concomitant hysterectomy or mesh type. At UNC, we reported on mesh exposure using a permanent suture for mesh attachment during SCP with and without concomitant total hysterectomy, with rates of 8% at 1 year.24 There is some evidence that a delayed absorbable suture may reduce the risk of mesh or suture erosion. In a retrospective review comparing braided permanent suture to delayed absorbable monofilament suture for SCP mesh attachment, rates of mesh exposure were reduced in the absorbable suture group (3.7% vs 0%), with no associated POP recurrence.25 Similarly, in another retrospective review, when delayed absorbable monofilament suture was used for SCP mesh attachment in 67 women undergoing total abdominal hysterectomy and SCP, no mesh exposures were noted at a median follow up of 27 months.26 The use of permanent sutures for vaginal mesh attachment has historically been advocated as a means to reduce POP recurrence risk; yet, no prospective study has definitively answered this question. The tradeoff of using a permanent suture may be an increased risk of mesh or suture exposure, as a permanent suture that has breached the vaginal epithelium may serve as a nidus for bacterial seeding, theoretically increasing the risk of mesh exposure. As SCP appears to be a more durable procedure for women with advanced uterovaginal prolapse, there is an urgent need to identify the ideal method of vaginal mesh attachment that minimizes the risk of mesh-related complications while maintaining effectiveness of the POP repair.

Choice of mesh material

Upsylon™ (Boston Scientific, Natick, MA) is a pre-formed Y-mesh that is light-weight (25 g/m2), composed of Type I polypropylene material, with a pore size of 2.8 mm2 and surface area ration of 1.11. It was FDA approved in 2012. The mesh is blue in color that may aide in the ability to detect even small areas of mesh exposure and erosion. No data currently exist regarding the performance of this particular mesh product in SCP. It is lighter in mesh weight than the IntePro™ y-mesh (American Medical Systems, Minneapolis, MN), which we previously used in the comparative trial of robotic to abdominal SCP in which our mesh exposure rates were 8%.

The primary aim of this randomized trial, therefore, is to test the hypothesis that use of the Upsylon™ mesh with a delayed absorbable suture for mesh attachment at the time of robotic-assisted total laparoscopic hysterectomy and SCP will reduce the risk of vaginal mesh and/or suture exposure compared to a permanent monofilament suture. Secondary aims will include an evaluation of the effect of this light-weight mesh and absorbable suture on prolapse and quality of life outcomes and surgical complications at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Subject must have apical with anterior or posterior vaginal prolapse with leading edge of prolapse to or beyond the hymen. This is defined as stage 2-4 pelvic organ prolapse ( C > - (TVL / 2) AND Ba or Bp ≥ 0 by the POP)
* Subject reports a bothersome bulge they can see or feel per PFDI-20, question 3, response of 2 or higher (i.e., responses of "somewhat", "moderately", or "quite a bit")
* Eligible for robotic or laparoscopic sacral colpopexy
* Desires surgical treatment for primary, symptomatic uterovaginal prolapse
* English speaking
* Willing to undergo hysterectomy

Exclusion Criteria:

* Patients who had prior hysterectomy
* Patients who are not surgical candidates due to medical comorbidities
* Current foreign body complications (including but not limited to erosion, fistula, abscess). This covers foreign bodies of any type (e.g. synthetic and biologic including allograft, xenograft).
* Desires uterine conservation
* Inability to give informed consent or to complete the testing or data collection
* Anticipated circumstances resulting in an inability to follow up (geographic relocation, etc).
* Pregnant or intends to become pregnant
* Active/chronic systemic infection including any gynecologic infection, untreated UTI or tissue necrosis
* History of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)
* Prior or currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Systemic connective tissue disease (e.g. scleroderma, Marfan's syndrome, Ehlers Danhlos, collagenosis, polymyositis or polymyalgia rheumatica)
* Chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Poorly controlled diabetes mellitus (DM), as indicated by Hemoglobin A1c > 9
* Those requiring concomitant rectopexy
* Subject is not able to conform to steep trendelenburg position
* Known sensitivity to polypropylene

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Geller, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Matthews CA, Geller EJ, Henley BR, Kenton K, Myers EM, Dieter AA, Parnell B, Lewicky-Gaupp C, Mueller MG, Wu JM. Permanent Compared With Absorbable Suture for Vaginal Mesh Fixation During Total Hysterectomy and Sacrocolpopexy: A Randomized Controlled Trial. Obstet Gynecol. 2020 Aug;136(2):355-364. doi: 10.1097/AOG.0000000000003884. PMID 32649494

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture
Started | 102 | 102
Surgery (Underwent sacral colpopexy) | 99 | 101
Completed (1 year follow-up) | 95 | 87
Not Completed | 7 | 15

BASELINE CHARACTERISTICS:
Population: The number of participants who underwent sacral colpopexy surgery
Groups:
- Total: Total of all reporting groups
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.7) | 59.0 (10.2) | 59.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 101 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 85 | 90 | 175
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 90 | 89 | 179
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 101 | 200
Current smoker [Count of Participants; unit: Participants] | 2 | 3 | 5
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (5.0) | 57.5 (4.7) | 27.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaginal Mesh or Suture Exposure
Description: Total number of participants with vaginal mesh and/or suture exposure thru 1 year
Time Frame: 1 year
Population: Participants who underwent sacral colpopexy surgery with 1-year follow up data
Measure: Count of Participants; unit: Participants
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture
Number analyzed (Participants) | 95 | 87
Participants | 5 | 8
Statistical Analysis 1: Comparison: Gore-Tex Permanent Suture vs PDS Delayed Absorbable Suture; Test type: Superiority; p = 0.30, Chi-squared; Risk Ratio (RR) = 1.74, 95% CI 2-sided [0.59 to 5.14]

2. Secondary Outcome: Number of Participants With Treatment Success
Description: Total number of participants with treatment success, which was a composite measure of 1) leading edge of prolapse not beyond hymen and apex not descended > 1/3 of vaginal length, 2) no subjective feeling of bulge on validated questionnaire, and 3) no prolapse re-treatment with pessary or surgery
Time Frame: 1 year
Population: Participants who underwent sacral colpopexy surgery with 1-year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture
Number analyzed (Participants) | 95 | 87
Participants | 88 | 83
Statistical Analysis 1: Comparison: Gore-Tex Permanent Suture vs PDS Delayed Absorbable Suture; Test type: Superiority; p = 0.43, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.96 to 1.11]

3. Secondary Outcome: Pelvic Floor Distress Inventory-20 (PFDI-20) Mean Score
Description: Condition-specific questionnaire, pelvic floor distress inventory-20 (PFDI-20) is used. Minimum value is 0. Maximum is 300. Higher scores mean more bothersome symptoms.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture
Number analyzed (Participants) | 95 | 87
score on a scale | 42.4 (35.9) | 37.9 (33.9)
Statistical Analysis 1: Comparison: Gore-Tex Permanent Suture vs PDS Delayed Absorbable Suture; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-14.7 to 5.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from surgery to 1 year follow-up visit, approximate total of 14 months
Description: Systematic assessment was performed with medical records review and detailed adverse event case report forms that were completed at study visits.
Arm/Group | Gore-Tex Permanent Suture | PDS Delayed Absorbable Suture
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 1/99 | 5/101
Other Adverse Events (participants affected / at risk) | 10/99 | 5/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gore-Tex Permanent Suture (N=99) | PDS Delayed Absorbable Suture (N=101)
Ureteral injury (Surgical and medical procedures) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Port site hernia (Surgical and medical procedures) | 0 (0) | 1 (1) — Port site hernia requiring surgery
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infected hematoma (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gore-Tex Permanent Suture (N=99) | PDS Delayed Absorbable Suture (N=101)
Intraoperative complications (Surgical and medical procedures) | 10 (10) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT02277925/Prot_SAP_000.pdf